CLINICAL TRIAL: NCT03664960
Title: A Phase 2, Multicenter, Open-Label, Extension Study to Evaluate the Safety and Tolerability of AK002 in Patients With Eosinophilic Gastritis and/or Eosinophilic Duodenitis (Formerly Referred to as Eosinophilic Gastroenteritis)
Brief Title: An Extension Study of AK002 in Patients With Eosinophilic Gastritis and/or Eosinophilic Duodenitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK002-003X
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Eosinophilic Gastritis; Eosinophilic Gastroenteritis; Eosinophilic Duodenitis
Keywords: Eosinophilic Gastritis; Eosinophilic Gastroenteritis; Eosinophil; EG; EGE; EGID; Eosinophilic gastrointestinal disorders; Eosinophilic Duodenitis; EoD
MeSH Terms: conditions — Eosinophilic enteropathy; Eosinophilic Esophagitis | interventions — AK002

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 to 3.0 mg/kg of AK002 (Experimental): Subjects in this arm will receive 26 monthly doses of AK002: a first dose of 1 mg/kg, followed by monthly doses of 3 mg/kg
  Interventions: Drug: AK002

INTERVENTIONS:
Drug: AK002 — AK002 is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8.

SUMMARY:
This is a Phase 2, open-label, extension study to assess the safety and tolerability of AK002, given monthly for up to 26 doses.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Completed Study AK002-003, defined as having received 4 infusions of study drug and followed through Day 113 (±3 days) in Study AK002-003 or discontinued from treatment due to high eosinophil counts prior to infusions 2, 3, or 4 and willing to begin extended dosing on or about Day 113 (for AK002-003 completers) or within 6 months of last dosing for patients discontinued from treatment.
3. If patient is on pre-existing dietary restrictions, willingness to note any changes that occur from the Baseline diet, throughout the study.
4. Able and willing to comply with all study procedures.
5. Female patients must be either post-menopausal for at least 1 year or surgically sterile (tubal ligation, hysterectomy, or bilateral oophorectomy) for at least 3 months, or if of childbearing potential, have a negative pregnancy test and agree to use dual methods of contraception, or abstain from sexual activity until the end of the study, or for 120 days following the last dose of study drug, whichever is longer.
6. Male patients with female partners of childbearing potential must agree to use a highly effective method of contraception until the end of the study or for 120 days following the last dose of study drug, whichever is longer. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant at any time during study participation.

Exclusion Criteria:

1. Poor tolerance to previous administration of AK002 in the opinion of the Investigator.
2. Known hypersensitivity to any constituent of the study drug.
3. Any disease, condition (medical or surgical), or cardiac abnormality, which, in the opinion of the Investigator, would place the patient at increased risk.
4. Vaccination with live attenuated vaccines within 30 days prior to initiation of treatment in the study, during the treatment period, or vaccination expected within 5 half-lives (4 months) of study drug administration. All types and formulations of vaccines (including live attenuated vaccines) authorized by FDA or other regulatory authority for the prevention of COVID-19 may be administered before, during, or after this study. The vaccine should not be administered within 7 days prior to and within 7 days after the administration of AK002 so that any side effects caused by either of the 2 medications can be more easily determined.
5. Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study.
6. Any other reason that, in the opinion of the Investigator or Medical Monitor, makes the patient unsuitable for enrollment.
7. Diagnosis of Hypereosinophilic Syndrome (HES), based on standard criteria (blood eosinophils >1500/µL with involvement of either the heart, nervous system, and/or bone marrow).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Paterson, MD, Study Director — Allakos Inc.
Locations (17):
- United States (17):
  - Phoenician Centers for Research and Innovation, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Ventura Clinical Trials, Ventura, California
  - Advanced Research Institute, New Port Richey, Florida
  - Northwestern, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - NIH, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - ClinSearch, Chattanooga, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Avant Research Associates, Austin, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants who were enrolled in and completed the study NCT03496571 had the option to participate in this open-label extension study.
Groups:
- Main Study Placebo to Extension Study 1 to 3.0 mg/kg of AK002: Subjects in this arm received the placebo in the main study (AK002-003) and were treated with 26 monthly doses of AK002: a first dose of 1 mg/kg, followed by monthly doses of 3 mg/kg.
  AK002: AK002 is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8.
- Main Study Active to Extension Study 1 to 3.0 mg/kg of AK002: Subjects in this arm received the active drug in the main study (AK002-003) and were treated with 26 monthly doses of AK002: a first dose of 1 mg/kg, followed by monthly doses of 3 mg/kg.
  AK002: AK002 is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8.
Period: Overall Study
Arm/Group | Main Study Placebo to Extension Study 1 to 3.0 mg/kg of AK002 | Main Study Active to Extension Study 1 to 3.0 mg/kg of AK002
Started | 21 | 37
Completed | 12 | 15
Not Completed | 9 | 22
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 3 | 14
Not completed — Sponsor Decision | 1 | 1
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study Placebo to Extension Study 1 to 3.0 mg/kg of AK002 | Main Study Active to Extension Study 1 to 3.0 mg/kg of AK002 | Total
Number analyzed (Participants) | 21 | 37 | 58
Age, Continuous [Median (Full Range); unit: years] | 35 [18 to 67] | 43 [18 to 74] | 40 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 26 | 35
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 21 | 32 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 21 | 33 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 37 | 58

OUTCOME MEASURES:

1. Primary Outcome: The Safety and Tolerability of AK002 by Evaluating Adverse Events Assessed Using the CTCAE Version 4.03
Description: Adverse events assessed using the CTCAE version 4.03
Time Frame: Through study completion, up to 28 months
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Placebo to Extension Study 1 to 3.0 mg/kg of AK002 | Main Study Active to Extension Study 1 to 3.0 mg/kg of AK002
Number analyzed (Participants) | 21 | 37
Participants
  Subjects with ≥1 adverse events | 21 | 35
  Subjects with ≥1 treatment-related adverse events | 15 | 22
  Subjects with an adverse event leading to study discontinuation | 0 | 3
  Subjects with ≥1 serious adverse events | 2 | 9
  Subjects with ≥1 treatment-related serious adverse events | 0 | 0

2. Secondary Outcome: Percent Change in PRO Total Symptom Score (TSS) From AK002-003 Baseline
Description: The PRO Total Symptom Score (TSS) is a patient-reported outcome (PRO) questionnaire comprises the following 8 symptoms: abdominal pain, nausea, vomiting, early satiety, loss of appetite, abdominal cramping, bloating, and diarrhea. Individual symptom scores ranged from 0 to 10. The daily total symptom score ranged from 0 to 80, with higher scores indicating greater severity. The End of treatment TSS score is defined as the average of the 14 daily scores on or after the day of the last dose of the extension study.
Time Frame: AK002-003 Baseline to End of Treatment (2 weeks post last dose, up to 26 months)
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Main Study Placebo to Extension Study 1 to 3.0 mg/kg of AK002 | Main Study Active to Extension Study 1 to 3.0 mg/kg of AK002
Number analyzed (Participants) | 21 | 37
Percentage of change | -66.3 (27.7) | -60.6 (32.4)

3. Secondary Outcome: Changes in the Number of Eosinophils in Gastric and/or Duodenal Mucosa From AK002-003 Baseline
Description: Percentage of Change in the Number of Eosinophils in Gastric and/or Duodenal Mucosa in each group from AK002-003 Baseline
Time Frame: AK002-003 Baseline to Day 547
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Main Study Placebo to Extension Study 1 to 3.0 mg/kg of AK002 | Main Study Active to Extension Study 1 to 3.0 mg/kg of AK002
Number analyzed (Participants) | 21 | 37
Percentage of change | -93.5 (18.9) | -99.7 (0.7)

ADVERSE EVENTS:
Time Frame: Through study completion, up to 28 months
Description: NCI Common Terminology Criteria for Adverse Events Version (CTCAE) 5.0 or most current version
Arm/Group | Main Study Placebo to Extension Study 1 to 3.0 mg/kg of AK002 | Main Study Active to Extension Study 1 to 3.0 mg/kg of AK002
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/37
Serious Adverse Events (participants affected / at risk) | 2/21 | 9/37
Other Adverse Events (participants affected / at risk) | 20/21 | 32/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study Placebo to Extension Study 1 to 3.0 mg/kg of AK002 (N=21) | Main Study Active to Extension Study 1 to 3.0 mg/kg of AK002 (N=37)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Abdominal hiernia (Gastrointestinal disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study Placebo to Extension Study 1 to 3.0 mg/kg of AK002 (N=21) | Main Study Active to Extension Study 1 to 3.0 mg/kg of AK002 (N=37)
Anemia (Blood and lymphatic system disorders) | 1 | 4
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2
Neutrophilia (Blood and lymphatic system disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 1 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 4 | 5
Vomiting (Gastrointestinal disorders) | 3 | 3
Chest pain (General disorders) | 1 | 3
Fatigue (General disorders) | 2 | 2
Influenza like illness (General disorders) | 2 | 1
Injection site pain (General disorders) | 3 | 1
Pyrexia (General disorders) | 2 | 1
Coronavirus infection (Infections and infestations) | 0 | 3
Influenza (Infections and infestations) | 2 | 4
Nasopharyngitis (Infections and infestations) | 5 | 5
Pneumonia (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 1 | 5
Urinary tract infection (Infections and infestations) | 1 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 9 | 11
Blood creatine phosphokinase increased (Investigations) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3
Headache (Nervous system disorders) | 3 | 7
Paresthesia (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 3 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement contains a limit on publication of results following completion of the trial. PIs are not allowed to publish results until a joint publication for the multicenter study or a set period of time. After that time, PIs may only publish results from their portion of the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT03664960/Prot_SAP_001.pdf